CLINICAL TRIAL: NCT02554760
Title: CoolSculpting the Flank Using an Applicator With a Crown Cooling Insert
Brief Title: Bilateral; Flank Study With Crown Cooling Insert
Acronym: CCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA15-004
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- All Study Participants (Experimental): This is a split body study in which all subjects will receive bilateral flank treatment with CoolSculpting. The investigator will determine one flank for treatment using the CoolCore applicator without an accessory for a duration of 60 minutes at a protocol-defined temperature. The contralateral flank will be treated with the standard CoolCore Applicator using an applicator accessory, the Crown Cooling Insert (CCI) at a protocol-defined temperature for a duration of up to 45 minutes. All enrolled subjects receive identical treatments; the investigator will use alternate subject numbers to balance which flank to treat with and without the CoolCore applicator accessory, such that all even subject numbers will receive treatment using the Standard CoolCore on the right flank and odd subject numbers will receive the same treatment on the left flank.
  Interventions: Device: The ZELTIQ CoolSculpting System

INTERVENTIONS:
Device: The ZELTIQ CoolSculpting System — The CoolSculpting device and CoolCore applicator with and without the Crown Cooling Insert will be used to perform the treatments.

SUMMARY:
Evaluate the safety and efficacy of non-invasive subcutaneous fat layer reduction in the flank using an applicator with and without the Crown Cooling Insert.

DETAILED DESCRIPTION:
This study will evaluate the Zeltiq CoolSculpting System when used with the standard CoolCore applicator and the CoolCore Applicator and the Crown Cooling Insert accessory.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects > 22 years of age and < 65 years of age.
* Subject has clearly visible fat on the flanks, which in the investigator's opinion, may benefit from the treatment.
* No weight change exceeding 5% of body weight in the preceding month.
* Subject with body mass index (BMI) up to 30. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
* Subject agrees to maintain his/her weight (i.e., within 5%) by not making any major changes in their diet or exercise routine during the course of the study.
* Subject has read and signed the study written informed consent form.

Exclusion Criteria

* Subject has had a surgical procedure(s) in the area of intended treatment.
* Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
* Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 12 months.
* Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
* Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Subject is taking or has taken diet pills or supplements within the past month.
* Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
* Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system
* Subject is pregnant or intending to become pregnant during the study period (in the next 5 months).
* Subject is lactating or has been lactating in the past 6 months.
* Subject has a history of hernia in the areas to be treated.
* Subject is unable or unwilling to comply with the study requirements.
* Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2015-12-17 (Actual); Study Completion 2015-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Kilmer, MD, Principal Investigator — Laser and Skin Surgery Center of Northern California
Locations (1):
- Laser and Skin Surgery of Northern California, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kilmer SL. Prototype CoolCup cryolipolysis applicator with over 40% reduced treatment time demonstrates equivalent safety and efficacy with greater patient preference. Lasers Surg Med. 2017 Jan;49(1):63-68. doi: 10.1002/lsm.22550. Epub 2016 Jun 21. PMID 27327898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects seeking a reduction in fat in the flank area were recruited from the general population.
Groups:
- Left Side With Crown Cooling Insert, Right Side Std CoolCore: Crown Cooling Insert (CCI) used for treatment on left flank at protocol-defined temperature and duration. Right flank treated using standard CoolCore applicator at protocol-defined temperature and duration.
- Left Side Std CoolCore, Right Side With Crown Cooling Insert: Left flank treated with standard CoolCore applicator at protocol-defined temperature and duration. Right side treated with Crown Cooling Insert at protocol-defined temperature and duration.
Period: Overall Study
Arm/Group | Left Side With Crown Cooling Insert, Right Side Std CoolCore | Left Side Std CoolCore, Right Side With Crown Cooling Insert
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CoolSculpting Treatment: The ZELTIQ CoolSculpting System: The CoolSculpting device and CoolCore applicator will be used to perform the treatments.
Arm/Group | CoolSculpting Treatment
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 46.7 [33 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 0
  Asian | 0
  Caucasian | 16
  Hispanic | 3
  Others | 0
Region of Enrollment [Number; unit: participants]
  United States | 19
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 25.3 [21 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Correctly Identified Pre-treatment Photos by a Panel of Blinded Independent Reviewers
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images of the treated areas. Reviewers will be practicing dermatologists or plastic surgeons. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images will be presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. Success will be defined as at least 70% correct identification of the pre-treatment images for flanks treated with each treatment parameter by at least 2 of 3 reviewers.
Time Frame: 12 weeks post-treatment
Population: All subjects received bilateral flank treatments.
Measure: Count of Units; unit: photos
Units Other Than Participants: photos
Groups:
- CoolSculpting Treatment With Standard CoolCore Applicator: 19 subjects received treatment for 60 minutes in duration at a protocol-defined temperature on one flank.
- CoolSculpting Treatment/ CoolCore Applicator Plus CCI: 19 subjects received treatment for a duration of 35 minutes at a protocol-defined temperature on the contralateral flank.
Arm/Group | CoolSculpting Treatment With Standard CoolCore Applicator | CoolSculpting Treatment/ CoolCore Applicator Plus CCI
Number analyzed (Participants) | 19 | 19
Number analyzed (photos) | 19 | 19
photos | 16 | 15
Statistical Analysis 1: Comparison: CoolSculpting Treatment With Standard CoolCore Applicator; Test type: Other; Catagorical tabulation; success proportion = 84.2, 95% CI 2-sided [60.4 to 92.3]
Statistical Analysis 2: Comparison: CoolSculpting Treatment/ CoolCore Applicator Plus CCI; Test type: Other; success proportion = 78.9, 95% CI 2-sided [54.4 to 93.9]

2. Primary Outcome: Safety of the Zeltiq CoolSculpting System Using the CoolCore Applicator With and Without the Crown Cooling Insert
Description: The safety endpoint is the number of unanticipated adverse device effects (UADE) as well as the number of device and/or procedure-related adverse events. Adverse events are collected from the time of enrollment through the 12 week final follow-up visit.
Time Frame: Enrollment through the 12 week post-treatment follow-up visit
Population: All 19 subjects were in the analysis group. Had there been any adverse events reported in the study period, each event would be categorized per intervention. However, there were zero adverse events reported for either of the two interventions and none reported for the study, therefore the arms were combined for the analysis.
Measure: Number; unit: UADEs /device or procedure events
Groups:
- CoolSculpting Treatment: The ZELTIQ CoolSculpting System: The CoolSculpting device and CoolCore applicator with and without the Crown Cooling Insert (CCI) will be used to perform the treatments.
  There were zero Unanticipated Adverse Device Events or device and/or procedure-related adverse events reported, therefore, both arms were aggregated for this analysis.
Arm/Group | CoolSculpting Treatment
Number analyzed (Participants) | 19
UADEs /device or procedure events | 0

3. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction as assessed by questionnaire administered at 12 weeks post-treatment. The questionnaire will consist of a 5-point Likert scale with the following selections options: 1) very unsatisfied; 2) somewhat unsatisfied; 3) neither satisfied nor unsatisfied; 4) somewhat satisfied; 5) very satisfied. jIn addition, free-text fields provided options for subjects responses.
Time Frame: 12 weeks post-treatment
Population: The per-protocol population (19 subjects) was included in the analysis. Each subject received treatment on each flank; the standard CoolCore applicator was used on one flank and the contralateral flank was treated with the CoolCore with the Crown Cooling Insert.
Measure: Count of Participants; unit: Participants
Groups:
- Standard CoolCore Without CCI: The CoolSculpting device and standard CoolCore applicator without the Crown Cooling Insert.
- Flank Treated With CoolCore + CCI: CoolCore Applicator with Crown Cooling Insert
Arm/Group | Standard CoolCore Without CCI | Flank Treated With CoolCore + CCI
Number analyzed (Participants) | 19 | 19
Participants
  Treatment was comfortable to very comfortable | 11 | 12
  Very visible to somewhat visible fat reduction | 10 | 10
  Satisfied to very satisfied with procedure | 13 | 12

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from enrollment through the 12-week post-treatment follow-up visit.
Description: There were no adverse events reported over the course of the study..
Groups:
- CoolSculpting Using Standard CoolCore: The CoolSculpting device using standard CoolCore applicator
- CoolSculpting Device Using Crown Cooling Insert: The CoolSculpting device using applicator and Crown Cooling Insert
Arm/Group | CoolSculpting Using Standard CoolCore | CoolSculpting Device Using Crown Cooling Insert
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No